CLINICAL TRIAL: NCT04176198
Title: A Phase 1/2, Open-Label, Dose-Escalation, Safety, Pharmacokinetic, and Pharmacodynamic Study of Oral Nuvisertib (TP-3654) in Patients With Intermediate or High-Risk Primary or Secondary Myelofibrosis
Brief Title: A Study of Oral Nuvisertib (TP-3654) in Patients With Myelofibrosis
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BBI-TP-3654-102
Record Dates: First submitted 2019-11-08; First posted 2019-11-25 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Myelofibrosis
MeSH Terms: conditions — Primary Myelofibrosis | interventions — TP 3654; ruxolitinib; N-(cyanomethyl)-4-(2-((4-(4-morpholinyl)phenyl)amino)-4-pyrimidinyl)benzamide

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm 1: nuvisertib (TP-3654) (Experimental)
  Interventions: Drug: Nusivertib
- Arm 2: nuvisertib (TP-3654) added on to ruxolitinib (Experimental)
  Interventions: Drug: Nusivertib; Drug: Ruxolitinib
- Arm 3: nuvisertib (TP-3654) in combination with momelotinib (Experimental)
  Interventions: Drug: Nusivertib; Drug: Momelotinib

INTERVENTIONS:
Drug: Nusivertib — Oral PIM Inhibitor
  Other Names: TP-3654
Drug: Ruxolitinib — Oral JAK inhibitor
  Other Names: Jakafi
  Arms: Arm 2: nuvisertib (TP-3654) added on to ruxolitinib
Drug: Momelotinib — Oral JAK inhibitor
  Other Names: Ojjaara
  Arms: Arm 3: nuvisertib (TP-3654) in combination with momelotinib

SUMMARY:
This study is a Phase 1/2, multicenter, dose-escalation, open-label trial to assess safety, tolerability, pharmacokinetics and pharmacodynamics of nuvisertib (TP-3654) in patients with intermediate or high-risk primary or secondary MF.

DETAILED DESCRIPTION:
Arm 1 will enroll patients who have been previously treated and failed on a JAK inhibitor or ineligible to receive treatment with a JAK inhibitor.

Arm 2 will enroll patients who are on a stable dose of ruxolitinib, but who have either lost response or had a suboptimal or plateau in response.

Arm 3 will enroll patients who have been previously treated with a JAK inhibitor (except momelotinib)

ELIGIBILITY:
Patients must meet all of the following inclusion criteria to be eligible:

Nuvisertib (TP-3654) Monotherapy Arm:

* Confirmed pathological diagnosis of primary myelofibrosis (PMF) or post-PV-MF/post-ET- MF and intermediate or high-risk primary or secondary MF
* Previously treated with JAK inhibitor(s) and is intolerant, resistant, refractory or has lost response to the JAK inhibitor(s) or is ineligible to be treated with JAK inhibitor
* Fulfill the following clinical laboratory parameters:
* Platelet count ≥ 25 x 10^9 /L, without assistance of growth factors or platelet transfusions
* ANC ≥ 1 x 10^9/L without assistance of granulocyte growth factors
* Peripheral blood blast count < 5%
* ECOG performance status ≤ 1
* Life expectancy ≥ 6 months
* Adequate renal function
* Adequate hepatic function
* Adequate coagulation function
* Splenomegaly (spleen volume of ≥ 450 cm3 by MRI or CT scan) within 2 weeks prior to Cycle 1 Day 1.
* Dose escalation: At least 2 symptoms measurable (score ≥ 1) using the MF-SAF
* Dose expansion: At least 2 symptoms measurable with each score of ≥ 3 or a total average score of ≥ 10 per MFSAF

Nuvisertib (TP-3654) + Ruxolitinib Arm:

* Confirmed pathological diagnosis of PMF or post-PV-MF/post ET- MF and intermediate or high-risk primary or secondary MF
* On ruxolitinib treatment for ≥ 6 months, and on a stable dose of ruxolitinib (5 to 25 mg BID) for ≥ 8 weeks prior to the first dose of nuvisertib, but has either lost response or had a suboptimal or plateau in response
* Fulfills the following clinical laboratory parameters:
* Platelet count ≥ 50 × 10^9/L (without assistance of growth factors or platelet transfusions)
* ANC ≥ 1 × 109/L without assistance of granulocyte growth factors
* Peripheral blood blast count < 5% at screening
* Adequate renal function
* Adequate hepatic function
* Adequate coagulation function
* Splenomegaly (spleen volume of ≥ 450 cm3 by MRI/CT scan) within 2 weeks prior to Cycle 1 Day 1
* At least 2 symptoms measurable with each score ≥ 3 or a total average score of ≥ 10 per MFSAF v4.0
* ECOG performance status ≤ 1
* Life expectancy ≥ 6 months

Nuvisertib (TP-3654) + Momelotinib Arm

* Confirmed pathological diagnosis of PMF or post-PV-MF/post ET-MF and intermediate or high-risk primary or secondary MF
* Previously treated with an approved JAK inhibitor (except momelotinib) for PMF or Post-PV/ET MF for ≥ 12 weeks, or ≥ 4 weeks if JAK inhibitor therapy was complicated by a transfusion requirement of ≥ 4 units of red blood cells in 8 weeks, or Grade 3/4 AEs of thrombocytopenia, anemia, or hematoma
* Fulfills the following clinical laboratory parameters:
* Anemic, defined as Hb <10 g/dL or requiring RBC transfusion at baseline
* Platelet count ≥ 50 × 109/L (without assistance of growth factors or platelet transfusions)
* ANC ≥ 1 × 109/L without assistance of granulocyte growth factors
* Peripheral blood blast count < 5% at screening
* Adequate renal function
* Adequate hepatic function
* Adequate coagulation function
* Splenomegaly (spleen volume of ≥ 450 cm3 by MRI/CT scan) within 2 weeks prior to Cycle 1 Day 1
* At least 2 symptoms measurable with each score of ≥ 3 or a total average score of ≥ 10 per MFSAF v4.0
* ECOG performance status ≤ 1
* Life expectancy ≥ 6 months

Patients meeting any one of these exclusion criteria will be prohibited from participating in this study:

Nuvisertib (TP-3654) Monotherapy Arm:

* Received previous systemic antineoplastic therapy or any experimental therapy within 2 weeks or 5 half-lives, whichever is longer, prior to Cycle 1 Day 1. Hydroxyurea or anagrelide are allowed up to 24 hours prior to Cycle 1 Day 1).
* Major surgery within 4 weeks prior to Cycle 1 Day 1 and/or not recovered adequately from from surgery prior to first dose.
* Splenic irradiation within 6 months prior to Screening or prior splenectomy.
* Prior allogeneic stem cell transplant within the last 6 months.
* Eligible for allogeneic bone marrow or stem cell transplantation.
* Unresolved Grade ≥ 2 non-hematological toxicity related to prior treatment
* History of symptomatic congestive heart failure, or myocardial infarction, or uncontrolled arrhythmia within 6 months prior to Cycle 1 Day 1; left ventricular ejection fraction (LVEF) < 45% by echocardiogram within 4 weeks prior to Cycle 1 Day 1.
* Corrected QT interval > 480msec.
* Prior or concurrent malignancy that could interfere with the investigational regime.
* Known history of chronic liver disease, e.g. portal hypertension or any of its complications, cirrhosis, Child-Pugh C, auto-immune hepatitis, alpha-1 anti-trypsin deficiency, Wilson's disease, etc.
* Active, uncontrolled bacterial, viral, or fungal infections, requiring systemic antimicrobial within 1 week prior to Cycle 1 Day 1.
* Chronic active or acute viral hepatitis A, B, or C infection (testing for hepatitis B and C are required)
* Exhibited allergic reactions or sensitivity to nuvisertib, or similar compound.
* Medical condition or GI tract surgery that could impair absorption or result in short bowel syndrome with diarrhea.
* Systemic steroid therapy (>10 mg daily prednisone or equivalent) within 1 week prior to the first dose of study treatment (note: topical, inhaled, nasal, and ophthalmic steroids are not prohibited).
* Known clinically significant anemia due to iron, vitamin B12, or folate deficiencies, or autoimmune or hereditary hemolytic anemia, or thalassemia, or severe GI bleeding.
* Pregnant or breastfeeding
* Currently receiving any other investigational agent.

Nuvisertib (TP-3654) + Ruxolitinib Arm:

* Received previous systemic antineoplastic therapy (other than ruxolitinib) or any other experimental therapy within 2 weeks or 5 half-lives, whichever is longer, prior to Cycle 1 Day 1 (Note: Prior treatment with nuvisertib is not allowed. Hydroxyurea or anagrelide are allowed up to 24 hours prior to Cycle 1 Day 1).
* Received systemic steroid therapy (>10 mg daily prednisone or equivalent) within 1 week prior to Cycle 1 Day 1 (Note: Topical, inhaled, nasal, and ophthalmic steroids are not prohibited)
* Known allergic reactions or sensitivity to nuvisertib, or similar compound.
* Splenic irradiation within 6 months prior to Screening or prior splenectomy
* Prior allogeneic stem cell transplant within the last 6 months (Note: Patients who have relapsed after 6 months post-transplant and do not have active GVHD are eligible).
* Eligible for allogeneic bone marrow or stem cell transplantation (Note: Patients who are not willing to undergo transplantation or for whom a suitable donor is not available are considered as transplant ineligible.)
* Major surgery within 4 weeks prior to Cycle 1 Day 1 and/or have not recovered adequately prior to first dose.
* Active, uncontrolled bacterial, viral, or fungal infections, requiring parenteral antimicrobial within 1 week prior to Cycle 1 Day 1
* Chronic active or acute viral hepatitis A, B, or C infection (testing for hepatitis B and C are required)
* Known history of chronic liver disease (eg, portal hypertension or any of its complications, cirrhosis, Child-Pugh C, auto-immune hepatitis, alpha-1 anti-trypsin deficiency, Wilson's disease, etc) (Note: Abnormal liver morphology at baseline imaging may require additional testing, as needed).
* Unresolved Grade ≥ 2 non-hematological adverse events related to prior treatment (stable Grade 2 conditions may be permitted in consultation with the Sponsor)
* History of myocardial infarction or symptomatic congestive heart failure or uncontrolled arrhythmia within 6 months prior to Cycle 1 Day 1; LVEF <45% by echocardiogram within 4 weeks prior to Cycle 1 Day 1
* Corrected QTcF of > 480 msec
* Prior or concurrent malignancy that could interfere with the safety or efficacy assessment of the study intervention
* History of a medical condition or GI tract surgery that could impair absorption or could result in short bowel syndrome with diarrhea
* Known clinically significant anemia due to iron, vitamin B12, or folate deficiencies, or autoimmune or hereditary hemolytic anemia, or thalassemia, or severe GI bleeding
* Pregnant or breastfeeding

Nuvisertib (TP-3654) + Momelotinib Arm:

* Received previous systemic antineoplastic therapy or any experimental therapy within 2 weeks or 5 half-lives, whichever is longer, prior to Cycle 1 Day 1 (Notes: Prior treatment with momelotinib or nuvisertib is not allowed; in patients with ongoing JAK inhibitor therapy, ie, ruxolitinib, at screening, JAK inhibitor therapy must be tapered over a period of at least 1 week. Patients on a low dose of ruxolitinib (eg, 5 mg QD) may have a reduced taper period or no taper; hydroxyurea or anagrelide are allowed up to 24 hours prior to Cycle 1 Day 1).
* Received systemic steroid therapy (>10 mg daily prednisone or equivalent) within 1 week prior to Cycle 1 Day 1 (Note: Topical, inhaled, nasal, and ophthalmic steroids are not prohibited).
* Known allergic reactions or sensitivity to nuvisertib, momelotinib, or any structurally similar drug, or to any component of the formulations of either study intervention
* Splenic irradiation within 6 months prior to screening or prior splenectomy
* Prior allogenic stem cell transplant within the last 6 months (Note: Patients who have relapsed after 6 months post-transplant and do not have active GVHD are eligible).
* Eligible for allogeneic bone marrow or stem cell transplantation (Note: Patients who are not willing to undergo transplantation or for whom a suitable donor is not available are considered as transplant ineligible).
* Major surgery within 4 weeks prior to Cycle 1 Day 1 and/or have not recovered adequately from surgery prior to first dose.
* Active, uncontrolled bacterial, viral, or fungal infections, requiring parenteral antimicrobial within 1 week prior to Cycle 1 Day 1
* Chronic active or acute viral hepatitis A, B, or C infection (testing for hepatitis B and C are required)
* Known history of chronic liver disease (eg, portal hypertension or any of its complications, cirrhosis, Child-Pugh C, auto-immune hepatitis, alpha-1 anti-trypsin deficiency, Wilson's disease, etc) (Note: Abnormal liver morphology at baseline imaging may require additional testing, as needed)
* Unresolved Grade ≥ 2 non-hematological adverse events related to prior treatment (stable Grade 2 conditions may be permitted in consultation with the Sponsor)
* Presence of Grade ≥ 2 peripheral neuropathy
* History of myocardial infarction or symptomatic congestive heart failure or uncontrolled arrhythmia within 6 months prior to Cycle 1 Day 1; LVEF < 45% by echocardiogram within 4 weeks prior to Cycle 1 Day 1
* Corrected QTcF of > 480 msec
* Prior or concurrent malignancy that could interfere with the safety or efficacy assessment of the study intervention
* History of a medical condition or GI tract surgery that could impair absorption or could result in short bowel syndrome with diarrhea
* Known clinically significant anemia due to iron, vitamin B12, or folate deficiencies, or autoimmune or hereditary hemolytic anemia, or thalassemia, or severe GI bleeding
* Pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2019-12-16 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2030-04-30 (Estimated)

PRIMARY OUTCOMES:
Determine the incidence of dose-limiting toxicities (DLTs) | 28 days
  Number of participants with DLTs
Determine the incidence of treatment emergent adverse events | From start of treatment to end of study
  Number of participants with Treatment Emergent Adverse Events and Serious Adverse Events
Assess patients for any evidence of preliminary activity by determining the number of patients with ≥ 35% spleen volume reduction (SVR35) | From start of treatment to end of study
  Number of participants with ≥ 35% spleen volume reduction (SVR35)

SECONDARY OUTCOMES:
Number of participants achieving objective response by IWG-MRT response criteria | From start of treatment to end of study
  Number of participants achieving complete remission, partial remission, clinical improvement, progressive disease and stable disease.
Number of participants who have ≥ 25% spleen volume reduction | Every 12 weeks from cycle 1 day 1 through cycle 19 day 1, and then every 24 weeks therafter during treatment.
  Number of participants who have ≥ 25% spleen volume reduction compared to baseline
Number of participants with ≥ 50% improvement in total symptom score (TSS50) at week 24 | 24 weeks
  Number of participants who have ≥ 50% total symptom score reduction by MFSAF compared to baseline after 24 weeks of treatment.
Determine the change in Patient Global Impression of Change (PGIC) at week 24 through end of study. | After 24 weeks of treatment to end of study
  Change in PGIC score
Determine the incidence of QT interval changes | 25 hours
  Changes in QT interval and heart rhythm
Establish the half-life (t½) of nuvisertib monotherapy, in combination with ruxolitinib, and in combination with momelotinib | 24 hours
  The estimate of time for the nuvisertib concentration or amount to be reduced by half
Establish the Area under the plasma concentration versus time curve (AUC) of nuvisertib monotherapy, in combination with ruxolitinib, and in combination with momelotinib | 24 hours
  The amount of drug exposure over 24 hours period after administration
Establish the Peak Plasma Concentration (Cmax) of nuvisertib monotherapy, in combination with ruxolitinib, and in combination with momelotinib | 24 hours
  The maximum nuvisertib concentration after administration
Establish the Time of Maximum concentration observed (tmax) of nuvisertib monotherapy, in combination with ruxolitinib, and in combination with momelotinib | 24 hours
  The time to reach maximum nuvisertib concentration

OTHER OUTCOMES:
Number of patients with reduction in bone marrow fibrosis | Every 24 weeks to end of study
Study potential pharmacodynamic (PD) markers of nuvisertib | 12 months
  Evaluate exploratory biomarkers, including change in protein phosphorylation and inflammatory cytokines, in peripheral blood samples and bone marrow biopsy samples.
Nuvisertib monotherapy: Changes in platelet count over time in patients with baseline platelet count < 100 x 10^9/L | From start of treatment to end of study
Nuvisertib combination arms: Assess the increase in hemoglobin ≥1.5 or ≥ 2 g/dL from baseline | From start of treatment to end of study
Nuvisertib combination arms: Assess red blood cell transfusion independence status or any requirement change | From start of treatment to end of study
Establish overall survival | From start of treatment to end of study
  The time interval from treatment start date to date of death from any cause

CONTACTS AND LOCATIONS:
Locations (80):
- United States (32):
  - University of Alabama, Birmingham, Alabama
  - The University of Arizona Cancer Center, Tucson, Arizona
  - City of Hope, Duarte, California
  - University of Southern California, Los Angeles, California
  - Hoag Family Cancer Institute, Newport Beach, California
  - Blood Cancer Center, Denver, Colorado
  - Yale School of Medicine, New Haven, Connecticut
  - University of Florida Health Shands Cancer Hospital, Gainesville, Florida
  - University of Miami, Miami, Florida
  - Baptist Health - Miami Cancer Institute, Miami, Florida
  - Emory University, Atlanta, Georgia
  - University of Chicago, Chicago, Illinois
  - University of Maryland, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Washington University of Medicine, St Louis, Missouri
  - John Theurer Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey
  - Roswell Park Comprehensive Cancer Center, Buffalo, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Weill Cornell Medical Center, New York, New York
  - Montefiore Cancer Center, The Bronx, New York
  - Duke Cancer Institute, Durham, North Carolina
  - Ohio State University, Columbus, Ohio
  - Medical University of South Carolina, Charleston, South Carolina
  - Tri-Star Centennial Medical Center, Nashville, Tennessee
  - Vanderbilt University, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - University of Washington - Fred Hutchinson Cancer Center, Seattle, Washington
- Australia (6):
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Eastern Health Box Hill Hospital, Box Hill, Victoria
  - Monash University, Clayton, Victoria
  - Peter McCallum Center, Melbourne, Victoria
  - Epworth Healthcare, Richmond, Victoria
  - Icon Cancer Centre (Ashford Cancer Centre Research), Adelaide
- Belgium (5):
  - University Hospitals Leuven, Leuven, Vlaams-Brabant
  - ZNA Cadix, Antwerp
  - ZNA Middelheim, Antwerp
  - Universitair Ziekenhuis Gent, Ghent
  - CHU de Liege, Liège
- Canada (5):
  - University of Calgary, Calgary, Alberta
  - St. Paul's Hospital Hematology/Oncology Research, Vancouver, British Columbia
  - University of British Columbia, Vancouver, British Columbia
  - Princess Margaret Cancer Center, Toronto, Ontario
  - Jewish General Hospital, Montreal, Quebec
- France (8):
  - Centre Hospitalier Universitaire D'Amiens, Amiens
  - CHU Angers, Angers
  - Centre Hospitalier Lyon Sud, Lyon
  - Hospitalier Universitaire (CHU) de Nice - Hopital de l'Archet, Nice
  - Institut de cancerologie du Gard, Nîmes
  - Hospital Saint Louis, Paris
  - University Hospital of Poitiers, Poitiers
  - Institut Gustave Roussy, Villejuif
- Italy (8):
  - Azienda Ospedaliera Nazionale SS. Antonio e Biagio e Cesare Arrigo, Alessandria
  - Istituto Nazionale Tumori, IRCCS Centro di Riferimento Oncologico di Aviano, Aviano
  - IRCCS Azienda Ospedaliero -Universitaria Di Bologna - Dipartimento Malattie Oncologiche ed Ematologiche - UO Ematologia, Bologna
  - ASST - Spedali Civili di Brescia, Brescia
  - IRCCS istituto Romagnolo per lo studio dei tumori "Dino Amadori", Meldola
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan
  - Università degli Studi di Milano-Bicocca, Milan
  - Azienda Ospedaliera Universitaria Citta' Della Salute E della Scienza di Torino, Torino
- Japan (12):
  - Aichi Medical University Hospital, Aichi
  - National Cancer Center Hospital East, Chiba
  - Kyushu University Hospital, Fukuoka
  - Hokkaido University Hospital, Hokkaido
  - University of Miyazaki Hospital, Miyazaki
  - Okayama University Hospital, Okayama
  - The University of Osaka Hospital, Osaka
  - Saitama Medical Center, Saitama
  - Tohoku University Hospital, Sendai
  - Shizuoka Cancer Center, Shizuoka
  - Juntendo University Hospital, Tokyo
  - Mie University Hospital, Tsu
- United Kingdom (4):
  - Lincoln County Hospital, Lincoln
  - United Lincolnshire Hospitals NHS Trust - Pilgrim Hospital, Lincoln
  - University College London Hospital's NHS foundation Trust, London
  - Oxford University Hospitals NHS Foundation, Oxford